CLINICAL TRIAL: NCT02050542
Title: Comparison of Prostate Cancer Detection Rates Obtained With Multiparametric MRI Targeted Transrectal Ultrasound Biopsies and Systematic Transrectal Ultrasound Biopsies.
Brief Title: Study of Current Practice Which Compare the Rate of Prostate Cancer by Using 2 Kind of Transrectal Biopsies: 3 by IRM-echography Image Fusion and 12 Systematized Guided Echographies.
Acronym: MURIELLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013-A00514-41; SC 3065 (Other: CPP)
Record Dates: First submitted 2014-01-29; First posted 2014-01-30 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: cancer; prostate; PSA; biopsies; ultrasound; MRI; fusion of images
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targeted biopsies guided by a fusion of MRI and ultrasound (Other): After the 12 systematic biopsies, the same patients will have to undergo 3 additional targeted biopsies on the suspicious image detected by IRM, guided by a fusion of MRI and ultrasound- images with the Koelis ® system
  Interventions: Procedure: systematic biopsies; Procedure: Targeted biopsies guided by a fusion of MRI and ultrasound- images
- Systematic biopsies (Other): The patients will have to undergo 12 systematic transrectal ultrasound-guided biopsies of the prostate
  Interventions: Procedure: systematic biopsies; Procedure: Targeted biopsies guided by a fusion of MRI and ultrasound- images

INTERVENTIONS:
Procedure: systematic biopsies — 90 patients will have to undergo 12 systematic transrectal ultrasound-guided biopsies of the prostate
  Other Names: Ultrasound-guided biopsies of the prostate
Procedure: Targeted biopsies guided by a fusion of MRI and ultrasound- images — Immediately after the 12 systematic biopsies, the same patients will have to undergo 3 additional targeted biopsies on the suspicious image detected by IRM, guided by a fusion of MRI and ultrasound- images with the Koelis ® system
  Other Names: Biopsies of the prostate by fusion of MRI and ultrasound- images with the Koelis ® system

SUMMARY:
The purpose of the study is to show that 3 targeted biopsies on the suspicious image detected by IRM, guided by a fusion of MRI and ultrasound- images with the Koelis ® system, will get no lower rate of cancer detection than those obtained by 12 systematic transrectal ultrasound-guided biopsies of the prostate.

DETAILED DESCRIPTION:
The act of current practice evaluated by this research is the act of prostate biopsies : the patient will have to undergo 12 systematized transrectal echography guided biopsies of the prostate and 3 additional biopsies targeted on the suspicious lesion detected with MRI, which are both done in current practice.

* A first operator is not informed of the location of the target. He will perform a series of 12 systematic transrectal ultrasound-guided biopsies of the prostate.
* Immediately after the second operator will perform 3 additional targeted biopsies on the suspicious image detected by IRM, guided by a fusion of MRI and ultrasound- images with the Koelis ® system

Act added by the research: Using a fusion of MRI - ultrasound images software system (Koelis ®).

ELIGIBILITY:
Inclusion Criteria:

* patient from 45 to 75 years old;
* Serum level of PSA > 4,0 ng / mL;
* Multiparametric prostate IRM, performed before inclusion and which confirm the diagnosis of suspected target;
* No opposition of the patient notified in the medical record
* patient member in a national insurance scheme.

Exclusion Criteria:

* Previous prostate biopsy;
* suspicious digital rectal examination;
* serum PSA > 20,0 ng / mL;
* treatment with 5 alpha reductase inhibitor during the last 3 months;
* untreated urinary infection

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Carcinomatous invasion on biopsies samples | Day 15
  The presence of carcinomatous invasion on biopsies samples

SECONDARY OUTCOMES:
Tissue length of biopsy invaded by the detected cancer | Day 15
  Maximal tissue length of biopsy invaded by the detected cancer
Biopsy Gleason score of the detected cancer | Day 15
  Maximal biopsy Gleason score of the detected cancer
Respective duration of each biopsy protocol | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: François Cornud, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (6):
- France (6):
  - CHU Grenoble, Grenoble
  - Chu Edouard Herriot, Lyon
  - CHU Pitié salpêtrière, Paris
  - CHU Cochin, Paris
  - CHU Toulouse Rangueil, Toulouse
  - Clinique Pasteur, Toulouse

REFERENCES:
- [Result] Delongchamps NB, Portalez D, Bruguiere E, Rouviere O, Malavaud B, Mozer P, Fiard G, Cornud F; MURIELLE Study Group. Are Magnetic Resonance Imaging-Transrectal Ultrasound Guided Targeted Biopsies Noninferior to Transrectal Ultrasound Guided Systematic Biopsies for the Detection of Prostate Cancer? J Urol. 2016 Oct;196(4):1069-75. doi: 10.1016/j.juro.2016.04.003. Epub 2016 Apr 12. PMID 27079582